CLINICAL TRIAL: NCT04319224
Title: An Open-label, Multi-center, Rollover Study in Subjects With Advanced Solid Tumor Malignancies After Participation in a Vopratelimab (JTX-2011) Clinical Study
Brief Title: Vopratelimab (JTX-2011) Alone and in Combination With Anti-Programmed Cell Death Protein 1 (PD-1) or Anti-Cytotoxic T-Lymphocyte Antigen 4 (CTLA-4) in Subjects With Advanced and/or Refractory Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to discontinue providing study drug to patients who have been on study treatment for more than two years
Sponsor: Jounce Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JTX-2011-R01
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: JTX-2011; Vopratelimab; Ipilimumab; Nivolumab; ICOS; Anti-CTLA-4; PD-1; PD-L1; Immunotherapy; Immuno-oncology; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vopratelimab (Experimental): Participants will continue to receive vopratelimab monotherapy per parent protocol.
  Interventions: Drug: Vopratelimab
- Vopratelimab with ipilimumab (Experimental): Participants will continue to receive vopratelimab in combination with ipilimumab per parent protocol.
  Interventions: Drug: Vopratelimab; Drug: Ipilimumab
- Vopratelimab with nivolumab (Experimental): Participants will continue to receive vopratelimab in combination with nivolumab per parent protocol.
  Interventions: Drug: Vopratelimab; Drug: Nivolumab

INTERVENTIONS:
Drug: Vopratelimab — Specified dose on specified days
  Other Names: JTX-2011
Drug: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy
  Arms: Vopratelimab with ipilimumab
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Vopratelimab with nivolumab

SUMMARY:
JTX-2011-R01 is an open label, multicenter, rollover study that is designed to provide continued access to vopratelimab for eligible subjects with advanced solid tumor malignancies who have previously participated in a vopratelimab study (the parent study).

DETAILED DESCRIPTION:
Vopratelimab is an agonist monoclonal antibody that specifically binds to the Inducible Co-Stimulator of T cells (ICOS) to generate an anti-tumor immune response. This is an open label, roll over study to evaluate the long-term safety of continued treatment with vopratelimab monotherapy or combination treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is currently receiving and tolerating vopratelimab (JTX-2011) therapy and receiving clinical benefit from study treatment in the opinion of the Investigator and/or Sponsor.
* Subject has demonstrated compliance with the parent study requirements, as assessed by the Investigator and/or Sponsor, and is able and willing to comply with the necessary visits and assessments as part of the rollover study.
* Written informed consent must be obtained prior to enrolling in the rollover study and receiving study treatment. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.
* Women of childbearing potential and males with partners of child-bearing potential must agree to use adequate birth control throughout their participation and for 5 months following the last study treatment

Exclusion Criteria:

* Subject was permanently discontinued from the parent study due to unacceptable toxicity, non-compliance with study procedures, withdrawal of consent, or any other reason.
* Subject is receiving concurrent anti-cancer treatment (excluding combination drugs such as nivolumab or ipilimumab as a component of the combination dosing regimen used in parent study).
* Women who are pregnant or breastfeeding.
* Subject has any medical or social condition that, in the opinion of the Investigator, might place a subject at increased risk, affect compliance, or confound safety or other clinical study data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stew Kroll, Study Director — Jounce Therapeutics, Inc.
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Health Systems, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vopratelimab: Participant received vopratelimab monotherapy (by intravenous infusion) at a dose of 0.1 mg/kg every 6 weeks
- Vopratelimab With Nivolumab: Participants received vopratelimab (by intravenous infusion) at a dose of 0.1 mg/kg or 0.3 mg/kg in combination with nivolumab (240 mg) every 3 weeks or every 6 weeks.
Period: Overall Study
Arm/Group | Vopratelimab | Vopratelimab With Nivolumab
Started | 1 | 3
Completed | 1 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vopratelimab | Vopratelimab With Nivolumab | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Adverse Events (AEs)
Description: Percentage of subjects with at least one AE
Time Frame: Approximately 34 months
Measure: Number; unit: percentage of participants
Arm/Group | Vopratelimab | Vopratelimab With Nivolumab
Number analyzed (Participants) | 1 | 3
percentage of participants | 100 | 100

2. Primary Outcome: Percentage of Subjects With Serious Adverse Events (SAEs)
Description: Percentage of subjects with at least one SAE
Time Frame: Approximately 34 months
Measure: Number; unit: percentage of participants
Arm/Group | Vopratelimab | Vopratelimab With Nivolumab
Number analyzed (Participants) | 1 | 3
percentage of participants | 100 | 0

3. Primary Outcome: Percentage of Subjects With Clinically Significant Change From Baseline in Clinical Laboratory Tests
Description: Percentage of subjects with at least one clinically significant change from baseline in clinical laboratory tests (i.e., change requiring adjustment of dose, clinical intervention or administration of concomitant medication)
Time Frame: Approximately 34 months
Measure: Number; unit: percentage of participants
Arm/Group | Vopratelimab | Vopratelimab With Nivolumab
Number analyzed (Participants) | 1 | 3
percentage of participants | 0 | 67

4. Secondary Outcome: Median Progression Free Survival (mPFS)
Description: mPFS from start of therapy on the rollover study (not including duration of treatment on the applicable parent study)
Time Frame: Approximately 34 months
Population: The PFS for the 1 participant receiving vopratelimab monotherapy and 2 of the 3 participants receiving vopratelimab in combination with nivolumab was censored due to non-occurrence of outcome event.
Measure: Median (Full Range); unit: months
Arm/Group | Vopratelimab | Vopratelimab With Nivolumab
Number analyzed (Participants) | 1 | 3
months | NA [NA to NA] — The PFS for the 1 participant in this arm/group was censored. | NA [9.8 to NA] — The PFS for 2 of the 3 participants in this arm/group were censored; therefore, no median was reached.

ADVERSE EVENTS:
Time Frame: Approximately 34 months
Groups:
- Vopratelimab With Nivolumab: Participants received vopratelimab (by intravenous infusion) at a dose of 0.1 mg/kg or 0.3 mg/kg in combination with nivolumab (240 mg) every 3weeks or every 6 weeks.
Arm/Group | Vopratelimab | Vopratelimab With Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vopratelimab (N=1) | Vopratelimab With Nivolumab (N=3)
Bladder transitional cell carcinoma (Renal and urinary disorders) | 1 (1) | 0 (0) — New primary malignancy: bladder transitional cell carcinoma
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vopratelimab (N=1) | Vopratelimab With Nivolumab (N=3)
Dry mouth (Gastrointestinal disorders) | 0 | 1 (1) — Grade 2
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 (1) — Grade 1
Pyrexia (General disorders) | 0 | 1 (1) — Grade 1
COVID-19 (Infections and infestations) | 0 | 2 (2) — Grade 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 (1) — Grade 2
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 — Grade 1
Papilloma viral infection (Infections and infestations) | 0 | 1 (1) — Grade 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 (1) — Grade 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 (2) — Grade 2
Alanine aminotransferase increased (Investigations) | 0 | 1 (1) — Grade 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 (1) — Grade 1
Neutrophil count decreased (Investigations) | 0 | 1 (1) — Grade 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 (3) — Grade 1
Headache (Nervous system disorders) | 0 | 1 (2) — Grade 1
Paraesthesia (Nervous system disorders) | 0 | 1 (1) — Grade 1
Anxiety (Psychiatric disorders) | 0 | 1 (1) — Grade 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) — Grade 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) — Grade 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 (1) — Grade 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 (1) — Grade 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 (1) — Grade 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1 (1) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT04319224/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04319224/SAP_001.pdf